CLINICAL TRIAL: NCT03095937
Title: Different Modalities for Evaluation of Fetal Cardiac Function in Pregnant Women With Rheumatic Heart Disease (RHD) Patients
Brief Title: Evaluation of Fetal Cardiac Function in Rheumatic Heart Disease (RHD) Patients
Acronym: RHD
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sief el eslam Ahmed Ali, Dr, Assiut University
Other Study IDs: ECHO001
Record Dates: First submitted 2017-03-20; First posted 2017-03-30 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Fetal Distress
MeSH Terms: conditions — Fetal Distress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to evaluate fetal myocardial performance in patients with heart diseases in comparison to normal pregnant patients.

DETAILED DESCRIPTION:
Cardiac diseases affect 1-4% of pregnancies of industrialized countries,and the number of patients who develop cardiac problems during pregnancy is increasing.

Congenital heart diseases, ischemic heart and cardiac arrhythmias are the most dominant causes. In developing countries, rheumatic heart disease remains prevalent. Pregnancy induces haemodynamic changes with increased intravascular volume which may not only poses a risk of maternal death but also of serious morbidity such as heart failure, stroke and cardiac arrhythmia.

The fetus is not spared.Previous reports revealed a significant reduction in fetal growth rates associated with maternal heart disease.There is also association with preterm delivery and reduced birth weight. The presence of maternal cyanosis and a reduced cardiac output are the most significant predictors.

Accurate and reliable measurement of fetal cardiac function could be valuable for making the diagnosis and for fetal surveillanceThe most suitable parameters for assessing fetal cardiac function will mainly be determined by the cause of the dysfunction. Abnormal values of ejection fraction or cardiac output are usually found in the late stages of deterioration, and therefore more sensitive parameters have been proposed for earlier diagnosis and monitoring of fetal cardiac dysfunction. In most cases of cardiac dysfunction, diastolic parameters (such as DV or IRT) are the first to be altered, reflecting impaired relaxation and compliance due to a stiffer or less effective heart. Similarly, parameters reflecting longitudinal function (such as annular displacement or velocities) are typically affected in the early stages as compared to radial function (such as ejection fraction).

The goal of this study is to evaluate fetal myocardial performance in patients with heart diseases in comparison to normal pregnant patients.

ELIGIBILITY:
Inclusion Criteria:

1. Compensated heart disease.
2. singleton pregnancy
3. Normal placental location
4. Have no associated hypertension, diabetes or any other medical disorders affecting pregnancy

Exclusion Criteria:

The patients have hypertension, diabetes or any other medical disorders affecting pregnancy.

Ages: 15 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pregnant women with compensated rheumatic heart disease and pregnant women with normal pregnancy with the same inclusion/exclusion criteria listed below.
  Inclusion criteria:
  1. Age of the patient: 15-40 years old.
  2. Compensated rheumatic heart disease.
  3. singleton Singleton pregnancy.
  4. Normal placental location.
  Exclusion criteria:
  The patients have hypertension, diabetes or any other medical disorders affecting pregnancy.
Sampling Method: Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Myocardial performance index | 30 minutes
  Percentage of isovolumetric time to ejection time

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided